CLINICAL TRIAL: NCT02573441
Title: KEYS to Succeed: Cognitive and Academic Intervention Program for Children and Adolescents Surviving Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Pediatric Oncology Group of Ontario (Other)
Responsible Party: Principal Investigator, Donald Mabbott, Program Head, Neurosciences & Mental Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000043747
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Childhood Brain Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Math + Liaison Service (Experimental): To help with mathematics, participants will be assigned to a workbook based version of the JUMP Math program which will be completed at home with a parent. This intervention focuses on mental math skills. In addition all participants will receive the liaison service program.
  Interventions: Behavioral: Jump Math; Behavioral: Liaison Services
- Working Memory + Liaison Service (Experimental): To help with working memory, participants will be assigned to Cogmed, a game-like computer exercise focusing on improving working memory. In addition all participants will receive the liaison service program.
  Interventions: Behavioral: Cogmed; Behavioral: Liaison Services
- Liaison Services (Other): Participants in this group will only receive the liaison service program for 12 weeks before being assigned to one of the intervention groups.
  Interventions: Behavioral: Liaison Services

INTERVENTIONS:
Behavioral: Jump Math — Jump Math is a workbook based program aimed at improving math skills
  Arms: Math + Liaison Service
Behavioral: Cogmed — Cogmed is an online computer program aimed at improving working memory skills
  Arms: Working Memory + Liaison Service
Behavioral: Liaison Services — Liaison Services will include working closely with schools to help explain the strengths and weaknesses of a child based on cognitive testing and to help with the implementation of recommendations

SUMMARY:
The study will examine whether school liaison services and home-based parental tutoring can help with academic difficulties of paediatric brain tumour survivors who received cranial spinal radiation and have returned to school. Forty-five patients will participate in the project. All patients will receive psychology liaison services to link resources at the hospital with those in the community. Patients will participate in one of two tutoring programs designed to directly or indirectly improve math skills over 12 weeks. Weekly phone calls will be used to support parents using the program. Patients will be tested before, immediately after, and six months following each tutoring program to assess growth in mathematics and working memory abilities.

DETAILED DESCRIPTION:
Paediatric brain tumour survivors who receive cranial spinal radiation have learning problems, particularly in mathematics and working memory. Working memory is often described as a "mental workspace" where relevant information is held in mind and processed. Working memory is important in mathematics for holding in mind relevant information and carrying out steps necessary to solve problems.

This study will examine whether school liaison support and home-based parental tutoring can help address the academic difficulties of paediatric brain tumour survivors who have received cranial spinal radiation and who have returned to their community school. Forty five patients will participate in the project. First, all patients will receive psychology liaison services to link resources at the hospital with those in the community in order to provide information regarding the effects of pediatric cancer on learning and facilitate the implementation of appropriate assistive technology and remediation programs. Patients will then participant in one of two tutoring programs over the course of a 12 week period. One group of patients will participate in a program that addresses working memory with the intent of indirectly helping with mathematics skills. This program will be delivered over the internet. Another group of patients will participate in a program using a work book to directly help improve mathematics skills. Weekly phone calls will be used to support parents in doing the program. Patients will be tested before, immediately after, and six months following each tutoring program to assess growth in mathematics and working memory abilities. The two intervention programs will be compared to a waitlist control group that receives only the liaison service (including academic support through weekly phone calls over the 12 weeks).

The findings from this study will provide evidence about the type of intervention that is most effective at helping paediatric brain tumour survivors improve their mathematics skills and working memory ability.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with a brain tumour and treated with cranial radiation
* Is between 1 and 10 years following diagnosis
* Has English as his or her native language or has had at least two years of schooling in English
* Is between the ages of 6 and 17
* Less than a Grade 8 equivalent math score

Exclusion Criteria:

* Is younger than 6 years or older than 17 years of age
* Is receiving palliative care

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Woodcock Johnson Academic-Third Edition | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of math Fluency, applied math problems, and qualitative concepts
Wechsler Intelligence Scale for Children - Fourth Edition Integrated | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of verbal and visual working memory
Wide Range Assessment of Memory and Learning - Second Edition | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of verbal and visual working memory
Automated Working Memory Assessment | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of verbal and visual working memory
Connors' Continuous Performance Test-Second Edition | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of sustained attention
Behaviour Rating Inventory of Executive Function-Parent Version | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of executive functioning
Monitoring Basic Skills Progress | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of mathematics

SECONDARY OUTCOMES:
SAM | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of participants attitude towards math
Wide Range Assessment of Memory and Learning - Second Edition | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of visual learning and memory
California Verbal Learning Test, Children's Version | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of verbal learning and memory
CANTAB | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  Measures of processing speed
Wechsler Abbreviated Scale of Intelligence - Second Edition | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  A measure of vocabulary and abstract visual reasoning
Delis-Kaplan Executive Function System | Pre-intervention, 12 weeks after intervention and 6 months follow-up
  Measures of processing speed and switching attention

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mabbott, Ph.D., Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada